CLINICAL TRIAL: NCT01089907
Title: Genomics Evolution in Childhood Acute Lymphoblastic Leukemia
Brief Title: Genomic Changes in Childhood Acute Lymphoblastic Leukemia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Lin Dong-Tsamn, National Taiwan University Hospital
Other Study IDs: 200906028R
Record Dates: First submitted 2010-03-17; First posted 2010-03-19 (Estimated); Last update posted 2010-03-19 (Estimated); Status verified 2010-03

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: genomic; childhood; acute lymphoblastic leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — bone marrow, peripheral blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To study the genomics with cell cycle and lymphocyte differentiation in disease, remission and relapse of childhood acute lymphoblastic leukemia. Then correlate these data with age, white cell count, cytogenetic changes, response to the chemotherapy and prognosis.

DETAILED DESCRIPTION:
In order to know the genomic evolution of childhood acute lymphoblastic leukemia, we will collect bone marrow (10c.c.) at diagnosis, remission and relapse. We will do the following genes in addition to gene-chip including IKZF1,ETV6, EBF1, NR3C1, RAG1/G2, TCF3, BTLA, PAX5,LEF1, ERG and VPREB1.We will study the gene dosages and degree of methylation. The estimated patients numbers will be 300-400. Then we will correlate these data with patients'age, white blood cell count at diagnosis, cytogenetic abnormalities, response to the chemotherapy and prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. patients diagnosed as acute lymphoblastic leukemia
2. age less than or equal to 18 years old
3. signed informed consent

Exclusion Criteria:

1. who is not acute lymphoblastic leukemia
2. who did not sign informed consent

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Acute lymphoblastic leukemia patients under 18 years of age
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2010-04; Primary Completion 2013-01 (Estimated); Study Completion 2013-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Tsamn Lin, M.D., Principal Investigator — National Taiwan University Hospital,Taipei,Taiwan
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan